CLINICAL TRIAL: NCT00752466
Title: A Drug Interaction Study of the Pharmacokinetics of Flunarizine and Topiramate (RWJ-17021-000) During Mono- and Concomitant Therapy
Brief Title: A Drug Interaction Study of the Pharmacokinetics of Topiramate and FLUNARIZINE When Given Together or Separately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Jan-Cil Italy (Unknown); Jan-Cil Spain (Unknown); Jan-Cil UK (Unknown); Jan-Cil Switzerland (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003283
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Human Volunteers; Migraine
Keywords: Healthy volunteers; drug interaction; Flunarizine; Topiramate; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; Flunarizine

INTERVENTIONS:
Drug: Topiramate; flunarizine

SUMMARY:
The primary purpose of this open-label study is to determine if concomitant therapy with topiramate and flunarizine has any effect on the pharmacokinetics of either drug. Safety will be assessed for all subjects, for the entire duration of the study.

DETAILED DESCRIPTION:
This is a multicenter, randomized open-label study to be conducted in 2 groups of subjects. Group 1 will consist of migraine patients to be recruited at multiple sites and Group 2 will include healthy subjects at a single study center. In Group 1 a total of 36 subjects will be enrolled with a target of having 24 subjects complete the study. In Group 2, a total of 28 healthy subjects will be enrolled so that at least 24 will complete the trial. Group 1 will include patients under treatment for migraine prophylaxis with any dose of flunarizine for at least 4 weeks prior to the 6-week run-in phase. Once selected, patients will enter a 6-week run-in phase in which they will receive 5mg of flunarizine every evening. Following this run-in phase, patients will continue on flunarizine and be randomized into 2 subgroups of equal size; Subgroup 1a will consist of patients being treated with topiramate and flunarizine and Subgroup 1b, the control group, where patients will only be receiving flunarizine treatment. Patients in Group 1 (Subgroups 1a and 1b) will commence initial confinement (Day 1) after completing the 6-week run-in phase. All these patients must have a history of migraine according to IHS1 criteria for at least 1 year prior to study entry. For both Groups 1 and 2 dropouts will be replaced to ensure the required number of patients/subjects of each sex to complete the study. Safety will be assessed by studying the incidence and severity of treatment-emergent adverse events and abnormal findings of other safety evaluations. Changes in clinical laboratory test and vital sign results from Baseline to End of Study or early termination will be evaluated.

In Group 1: 5 mg flunarizine every 24 hours (at 8:00 p.m.), beginning on Day -42 for 6 weeks, through Day -1. Patients will continue to receive this dose from Days 1 through 81. Group 1a: On Day 4 Topiramate dose titrated from 25 mg BID to 75 mg (25 mg am and 50 mg pm) by Day 19 and 50 mg BID by Day 26 - Day 81. Group 1b continue on Flunarizine only. Group 2: Topiramate beginning Day 2 titration from 25 mg BID to 50 mg BID by Day 5 through 18. 5mg Flunarizine daily starting Day 12- Day 18.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in Group 1 must be diagnosed with migraine for at least 1 year prior to study start. Subjects must also have received any dose of flunarizine for the prophylaxis of migraine, for a minimum of 4 weeks prior to the run-in phase. Subjects in Group 2 must be healthy subjects
* Weight within 15% of the ideal body weight according to height and frame size
* Healthy based on a detailed medical history, physical examination, and clinical laboratory evaluations
* Normal ECG at the time of screening
* Women of non-child bearing potential or practicing acceptable birth control
* Negative pregnancy test within 4 days of run-in phase
* Signed informed consent

Exclusion Criteria:

* History of significant medical disease (e.g., ophthalmologic, cardiovascular, renal, hepatic, gastrointestinal, hematological, endocrine, metabolic, neurologic or psychiatric disease)
* Conditions known to be contraindications to the use of flunarizine including obesity, hypotension, a history of depressive illness or pre-existing symptoms of Parkinson's disease or other extrapyramidal disorders
* History of an acquired or hereditary neurologic disease, e.g., epilepsy or significant brain trauma
* Subjects who are schizophrenic, exhibit bipolar disorder, or have exhibited any psychotic symptoms or have a history of any serious psychiatric disorder, including suicide attempt
* Subjects demonstrating significant active physical disease, acute or chronic, within 7 days prior to the start of the study
* Active liver disease
* Clinically significant abnormal laboratory tests including, but not limited to, an out-of-range screening TSH level, LFT levels greater than or equal to 2 times above the upper limit of normal, a creatinine level above the upper limit of normal
* Personal or family history of nephrolithiasis
* Allergy to heparin
* History of drug allergy or hypersensitivity to sulfonamides (including RWJ-17021-000, topiramate)
* Malignancy or history of malignancy within the last 5 years with the exception of treated basal cell carcinoma
* Glaucoma
* Testing positive for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, and drugs of abuse, including alcohol
* History of alcohol or drug abuse
* Subjects taking concomitant medications within 14 days prior to Day 1 including iodinated contrast materials that have not been preapproved by the Medical Monitor and Global Clinical Pharmacokinetics Leader
* Subjects who have taken medications that are known cytochrome P450 inducers or inhibitors (see Attachment 4) within the 28 days prior to Day 1
* Subjects who have taken prescription medications within 14 days prior to Day 1 (with the exception of chronic thyroid therapy and rescue/abortive medication for migraine headache) or
* Over-the-counter medications (including aspirin, vitamins) within 7 days prior to Day 1 or antacids within the 48 hours prior to Day 1
* Use tobacco products during the 3 months prior to screening
* Consumption of grapefruit and Seville orange containing products, or herbal medications within the 28 days prior to Day 1
* Drinking alcohol for at least 7 days prior to Day 1
* Subjects who have not limited the consumption of methylxanthine containing products to 2, 8 oz. drinks/day or less within the 24 hours prior to each confinement
* Female subjects who are pregnant and/or nursing
* Subjects who have received an experimental drug, donated blood, or used an experimental medical device within 30 days prior to screening (also subjects who have been recent participants in a topiramate study, within 2 weeks of screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2003-03; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
For each treatment and each group, the plasma concentration at each time point and the pharmacokinetic parameters of interest will be summarized using descriptive summary statistics.

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events and abnormal findings of other safety evaluations. Changes in clinical laboratory test and vital sign results from Baseline to End of Study or early termination will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Drug Interaction Study of the Pharmacokinetics of Flunarizine and Topiramate (RWJ 17021 000) During Mono- and Concomitant Therapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=519&filename=CR003283_CSR.pdf